CLINICAL TRIAL: NCT05486728
Title: A Double-Blinded, Parallel, Vehicle-Controlled Phase 2 Study of SHJ002 Sterile Ophthalmic Solution in Participants With Dry Eye Disease
Brief Title: Phase II Study of SHJ002 Sterile Ophthalmic Solution Compared With Vehicle in Participants With Dry Eye Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dreamhawk Vision Biotech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SHJ002-DED2203
Record Dates: First submitted 2022-08-02; First posted 2022-08-04 (Actual); Results first posted 2025-10-14 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-09

CONDITIONS: Dry Eye Disease
Keywords: Dry Eye Disease
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Intervention Model Description: Double-Blinded, Parallel, Vehicle-Controlled
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SHJ002 (Experimental): SHJ002 Ophthalmic Solution: topically administered to each eye BID for 84 days
  Interventions: Drug: SHJ002/Vehicle
- Vehicle (Placebo Comparator): Vehicle: topically administered to each eye BID for 84 days
  Interventions: Drug: SHJ002/Vehicle

INTERVENTIONS:
Drug: SHJ002/Vehicle — Topical ophthalmic

SUMMARY:
The purpose of this study is to measure efficacy and safety with SHJ002 sterile ophthalmic solution compared to vehicle in participants with Dry Eye Disease (DED). SHJ002 is an antisense oligonucleotide to neutralize a specific microRNA.

DETAILED DESCRIPTION:
Participants will be randomized to treatment with SHJ002 Ophthalmic Solution or vehicle which will be administered to each eye BID for 84 days.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants 18 years of age or older inclusive, at the time of signing the informed consent.
2. Have DED in both eyes for ≥ 6 months
3. Female participants must be 1 year postmenopausal, surgically sterilized, or females of childbearing potential with a negative urine pregnancy test

Exclusion Criteria:

1. Ocular surface corneal disease, other than DED.
2. Lid margin disorder other than meibomian gland dysfunction (MGD)
3. Presence of any ocular condition
4. Any history of eyelid surgery or intraocular/ocular surgery
5. Cauterization of the punctum or punctal plug
6. Use of lid scrubs containing chemicals or baby shampoo, or eye makeup
7. Use of any of the contraindicated drugs medications
8. Any changes in the dosing of any chronically used systemic drug
9. Disease, condition, or disorder that in the judgement of Investigator could confound study assessments or limit compliance to study protocol
10. Known history of alcohol and/or drug abuse within 12 months
11. Known allergy or contraindication to any component of investigational product (IP) formulation or diagnostic agents.
12. Participation in any drug or device clinical investigation within 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2023-02-08 (Actual); Primary Completion 2023-12-07 (Actual); Study Completion 2023-12-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- Australian Eye Specialists, Werribee, Victoria, Australia
- Kaohsiung Veterans General Hospital, Kaohsiung City, Kaohsiung, Taiwan
- Thailand (2):
  - King Chulalongkorn Memorial Hospital, Bangkok
  - Ramathibodi Hospital, Mahidol University, Bangkok

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | SHJ002 | Vehicle
Started | 42 | 43
Completed | 42 | 41
Not Completed | 0 | 2

BASELINE CHARACTERISTICS:
Population: FAS population
Groups:
- Total: Total of all reporting groups
Arm/Group | SHJ002 | Vehicle | Total
Number analyzed (Participants) | 42 | 43 | 85
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.9 (15.08) | 45.7 (14.28) | 46.3 (14.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 32 | 61
  Male | 13 | 11 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 42 | 42 | 84
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 40 | 42 | 82
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 2 | 1 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Weight [Mean (Standard Deviation); unit: kg] | 64.30 (10.820) | 63.80 (12.990) | 64.10 (11.900)
Height [Mean (Standard Deviation); unit: cm] | 161.2 (7.77) | 159.7 (8.42) | 160.5 (8.10)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Total Corneal Fluorescein Staining (NEI Scale)
Description: NEI Corneal Fluorescein Staining Score (range: 0 to 15, where higher scores indicate worse corneal staining). The score is the sum across five corneal regions (each 0-3).
Time Frame: Baseline and Day 84
Population: FAS population
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | SHJ002 | Vehicle
Number analyzed (Participants) | 42 | 43
score on a scale | -2.4 [-3.08 to -1.69] | -1.3 [-2.03 to -0.64]

2. Secondary Outcome: Change From Baseline in SANDE Score
Description: The SANDE questionnaire assesses dry eye symptoms on a scale from 0 (no symptoms) to 100 (worst symptoms). The reported values represent change from baseline to Day 84 (Day 84 - Baseline).
Time Frame: Baseline and Day 84
Population: FAS population
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | SHJ002 | Vehicle
Number analyzed (Participants) | 42 | 43
score on a scale | -43.9 [-49.48 to -38.3] | -36.0 [-41.71 to -30.39]

3. Secondary Outcome: Change From Baseline in Eye Dryness Score (Visual Analogue Scale)
Description: 100-mm horizontal line from 0 (no discomfort) to 100 (worst discomfort). Reported values represent change from baseline to Day 84.
Time Frame: Baseline and Day 84
Population: FAS population
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | SHJ002 | Vehicle
Number analyzed (Participants) | 42 | 43
score on a scale | -32.0 [-38.03 to -25.89] | -23.3 [-29.08 to -17.42]

ADVERSE EVENTS:
Time Frame: 84 days
Arm/Group | SHJ002 | Vehicle
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/43
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/43
Other Adverse Events (participants affected / at risk) | 0/42 | 0/43

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-07-07): https://cdn.clinicaltrials.gov/large-docs/28/NCT05486728/Prot_SAP_000.pdf